CLINICAL TRIAL: NCT04986137
Title: Diagnostic Performance of Fractional Excretion of Urea in Acute Kidney Injury in Patients With Liver Cirrhosis
Brief Title: Fractional Excretion of Urea for the Differential Diagnosis of Acute Kidney Injury in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Khalaf Mahmoud, Assistant lecturer of Internal Medicine. Faculty of Medicine, Aswan University, Sohag University
Other Study IDs: Soh-Med-21-07-25
Record Dates: First submitted 2021-07-16; First posted 2021-08-02 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Injury
Keywords: ascites; hepatorenal syndrome; acute tubular necrosis; pre-renal azotemia; cirrhosis
MeSH Terms: conditions — Acute Kidney Injury; Ascites; Hepatorenal Syndrome; Kidney Cortex Necrosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Acute kidney injury due to acute tubular necrosis
- Group 2: Acute kidney injury due to prerenal azotemia
- Group 3: Acute kidney injury due to hepatorenal syndrome type 1

SUMMARY:
The aim of this study is to evaluate:

* The diagnostic performance of Fractional Excretion of Urea (FEUrea) for the differential diagnosis of acute kidney injury in patients with cirrhosis and ascites presenting to a tertiary care hospital.
* The ability of Fractional Excretion of Urea to distinguish between

  1. structural group of acute kidney injury (acute tubular necrosis) versus functional group of acute kidney injury (prerenal azotemia and hepatorenal syndrome), and
  2. types of functional group (prerenal azotemia versus hepatorenal syndrome type 1).

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication of end-stage liver disease and is one of the criteria that define acute-on-chronic liver failure.

There are two types of AKI in cirrhosis: functional and structural. The functional group is divided into the volume responsive prerenal azotemia (PRA) that results from decreases in intravascular volume (e.g., aggressive diuretic treatment, diarrhea) and volume-unresponsive state or called hepatorenal syndrome (HRS). AKI that is unresponsive to albumin infusion and withdrawal of diuretics in the absence of identifiable causes. The structural group includes acute tubular necrosis (ATN) that results from intrinsic damage and other renal parenchymal disorders.

Urea is filtered in the glomerulus and then largely reabsorbed in the proximal tubule and also in the distal tubule. The reabsorption of urea is increased by vasopressin and the renin-angiotensin-aldosterone system. The fractional excretion of urea under conditions of decreased renal perfusion and increased vasopressin and renin-angiotensin-aldosterone system (RAAS), such as that seen in cirrhosis with PRA or HRS type 1, should therefore decrease. Conversely, renal tubular injury should impair reabsorption and increase its fractional excretion. Since urea absorption is largely modulated in the proximal tubules, it is not affected by diuretics acting more distally. Recently it is therefore hypothesized that the fractional excretion of urea (FEUrea) could serve as a clinical aid in making an early distinction between ATN versus PRA and HRS type 1 in patients with cirrhosis and ascites presenting with AKI. The current study was designed to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years.
* Decompensated liver cirrhosis (Child-Pugh classification B or more) of any etiology diagnosed by clinical parameters involving laboratory tests, endoscopic or radiologic evidence of cirrhosis, history of decompensation (hepatic encephalopathy, ascites, variceal bleeding, jaundice), and liver biopsy if available.
* Use of either loop diuretics and/or distal diuretics (ex; spironolactone and eplerenone) until the time of admission.
* Availability of a baseline serum creatinine as defined by the International Club Ascites.

Exclusion Criteria:

* Prior liver or kidney transplant
* Advanced chronic kidney disease defined as serum creatinine greater than 4 mg/dL
* Patients on acute or chronic renal replacement therapy
* Patients with hepatocellular carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential patients will be identified by screening all cirrhotic patients who will be admitted with acute kidney injury to a specialized hepatology inpatient unit or who will attend for follow up at outpatient clinics
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in fractional excretion of urea percentage in urine | "through study completion, an average of 1 year".
  By equation : [(urine Na ÷ serum Na) ÷ (urine creatinine ÷ serum creatinine)] x 100%

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Sabet, Professor, Principal Investigator — Suhag University
Locations (1):
- Aswan University Hospitals, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No